CLINICAL TRIAL: NCT02370953
Title: VERION Versus Conventional, Manual Ink-marking in Toric IOL Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL51895.068.14
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2015-11

CONDITIONS: Astigmatism
Keywords: Toric IOL alignment; VERION digital marker; Manual ink-marking; Randomized controlled trial
MeSH Terms: conditions — Astigmatism | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VERION (Experimental): In this group the VERION-tools (Digital Marker) are used for the alignment of the toric IOL
  Interventions: Device: VERION for toric IOL alignment
- Conventional, manual ink-marking (Active Comparator): In the group the conventional manual marking is used for the alignment of the toric IOL
  Interventions: Procedure: Conventional, manual ink-marking for toric IOL alignment

INTERVENTIONS:
Device: VERION for toric IOL alignment — The VERION Measurement Module is a diagnostic device which can make high resolution colour reference images of the patient's eye for position reference. The VERION Digital Marker is a medical device that assists the surgeon in planning and performing surgical procedures on the eye. The VERION tools use several reference points on the conjunctiva and limbus, and make an overlay between the preoperative achieved and live-surgery image. During surgery, this device projects the horizontal axis and the estimated placement axis of the toric IOL on the patient's eye, and therefore, the surgeon can accurately place the toric IOL to its preoperatively calculated angle.
  Other Names: VERION Measurement Module and Digital Marker
  Arms: VERION
Procedure: Conventional, manual ink-marking for toric IOL alignment — Several manually performed methods are used to align the toric IOL at the intended axis. Most of them use a 3-step procedure. First, the horizontal axis of the eye is temporarily marked with ink in a seated position to correct for cyclotorsion when changing into supine position. Three spots on the conjunctiva, close to the edge of the cornea, are applied at 0°, 90° and 180°, which may be done by using a bubblemarker or gravity marker with a calibrated horizontal position. Next, the desired alignment axis for the toric IOL is marked intra-operatively. The last step is to rotate the implanted toric IOL until the IOL markings agree with the alignment marks. After surgery is performed, the ink marks will disappear within a few hours.
  Other Names: Conventional, manual ink-marking
  Arms: Conventional, manual ink-marking

SUMMARY:
OVERVIEW Cataract is a clouding of the crystalline lens which causes vision loss and blindness if untreated. Cataract surgery is the most frequently performed surgical intervention in medicine with an incidence of 880 surgeries per 100.000 population in 2010 amounting to a total number of over 160.000 surgeries per year in the Netherlands.

Approximately 22% of patients with cataract have a substantial pre-existing corneal astigmatism. Toric IOLs provide the opportunity to correct pre-existing astigmatism, offering the patients optimum distance vision without the use of spectacles or contact lenses. Toric IOLs are increasingly used in cataract and refractive surgery.

Since the introduction of toric intraocular lenses (IOLs) in the treatment of cataract in patients with pre-existing corneal astigmatism, numerous studies have shown the importance of accurate positioning of the toric IOL to the intended alignment axis. An error of 5º in toric IOL alignment will decrease the anticipated effect by 17% and thus misalignment will decrease the effectiveness of the astigmatism treatment. There are several methods used to align the toric IOL at the intended axis. Most of these use a 3-step ink-marking procedure and are performed manually. Clinical study showed an average error of 5º in toric IOL alignment when using this method.

Two new tools that have recently been introduced to the market are the VERION Measurement Module and VERION Digital Marker. Together, these tools provide integrated digital guidance for alignment of toric IOLs and they have the potential to eliminate the error in horizontal axis marking and the alignment axis marking error. This will lead to an improved visual outcome. So far, there are no published studies using the VERION tools for toric IOL alignment in cataract surgery. Therefore, the investigators will perform this randomized control trial.

MAIN HYPOTHESIS

The investigators hypothesise that cataract surgery with the implantation of a toric IOL, when using the VERION-tools, compared to manual ink-marking, in patients with corneal astigmatism will lead to:

- An increase in accuracy in toric IOL alignment

OBJECTIVES

Primary Objective:

The primary objective of the study is to compare the accuracy in toric IOL alignment when using the VERION-tools for alignment of the toric IOL or the conventional manual ink-marking procedure.

Other hypotheses and objectives are available in the detailed description.

DETAILED DESCRIPTION:
Extra hypotheses

* A decrease in residual astigmatism
* An improved best corrected distance visual acuity (BCVA)
* An improved uncorrected distance visual acuity (UCVA)
* A decrease in residual refractive astigmatism
* A decrease or comparable complication profile

Secondary Objective:

The secondary objective of the study is to compare residual astigmatism when using the VERION Measurement Module and VERION Digital Marker for alignment of the toric IOL or the conventional manual ink-marking procedure.

Other Secondary Objectives:

The other secondary objectives are to compare:

1. Best corrected distance visual acuity (BCVA)
2. Uncorrected distance visual acuity (UCVA)
3. Residual refractive astigmatism
4. Wavefront aberrations
5. Complication profile

ELIGIBILITY:
Inclusion Criteria:

* Astigmatism (at least 1.25D)
* Cataract
* Are at least 18 years of age
* Eye eligible to undergo cataract extraction
* Eye eligible for toric IOL implantation
* Bilateral eyes: availability to undergo second eye surgery within 2 weeks of the first eye surgery
* Willing and able to comply with scheduled visits and other study procedures
* Understand and signed informed consent

Exclusion Criteria:

* Irregular corneal astigmatism or keratoconus
* Extensive age related macular degeneration (atrophic or exudative AMD or numerous soft drusen)
* Fuchs endothelial dystrophy (stage 2)
* Uncontrolled/manifest glaucoma
* Glaucoma related extensive visual field loss
* Extensive diabetic macular disease
* Previous intraocular or corneal surgery of any kind
* Subjects presenting any contraindications to cataract surgery
* Subjects with a recurrent or active ocular or uncontrolled eyelid disease
* Subjects with a history of lens instability (e.g. posterior polar cataract, traumatic cataract) or zonular instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Average error (in degrees) in toric IOL-axis | at week 13 (after the first surgery, if bilateral surgery was performed).

SECONDARY OUTCOMES:
Percentage of eyes with residual refractive cylinder ≤0.5D | at week 13 (after the first surgery, if bilateral surgery was performed).

OTHER OUTCOMES:
Best corrected distance visual acuity (BCVA) | at week 13 (after the first surgery, if bilateral surgery was performed).
Uncorrected distance visual acuity (UCVA) | at week 13 (after the first surgery, if bilateral surgery was performed).
Residual refractive astigmatism | at week 13 (after the first surgery, if bilateral surgery was performed).
Complication profile | at week 13 (after the first surgery, if bilateral surgery was performed).

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Nuijts, MD, PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Bauer NJ, de Vries NE, Webers CA, Hendrikse F, Nuijts RM. Astigmatism management in cataract surgery with the AcrySof toric intraocular lens. J Cataract Refract Surg. 2008 Sep;34(9):1483-8. doi: 10.1016/j.jcrs.2008.05.031. PMID 18721707
- [Result] Visser N, Berendschot TT, Bauer NJ, Jurich J, Kersting O, Nuijts RM. Accuracy of toric intraocular lens implantation in cataract and refractive surgery. J Cataract Refract Surg. 2011 Aug;37(8):1394-402. doi: 10.1016/j.jcrs.2011.02.024. PMID 21782085
- [Result] Visser N, Berendschot TT, Verbakel F, de Brabander J, Nuijts RM. Comparability and repeatability of corneal astigmatism measurements using different measurement technologies. J Cataract Refract Surg. 2012 Oct;38(10):1764-70. doi: 10.1016/j.jcrs.2012.05.036. PMID 22999600